CLINICAL TRIAL: NCT04371120
Title: Brain Injury Self-Efficacy Scale Validation
Acronym: BICSQ
Status: Terminated | Type: Observational
Why Stopped: Funding
Sponsor: Rehabilitation Hospital of Indiana (Other)
Responsible Party: Sponsor
Other Study IDs: 1902472436
Record Dates: First submitted 2019-08-08; First posted 2020-05-01 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury; Self Efficacy
Keywords: Traumatic Brain Injury; Self Efficacy; Validation
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brain Injury Survivors: Traumatic or acquired brain injury survivors, patients of RHI
  Interventions: Diagnostic Test: BICS Q

INTERVENTIONS:
Diagnostic Test: BICS Q — assess perceived self-efficacy (PSE) regarding a person's brain injury and proved responsive to treatment effects in the original BICS study.15-16 Specifically, it measures a person's perceptions about his or her ability to both understand the effects of brain injury, as well as, perceived capability of managing BI-related challenges. As the literature suggests, it is important to utilize a measure that would assess PSE specific to the person's challenge, rather than a general PSE scale.

SUMMARY:
The purpose of this study is to validate the Brain Injury Self-Efficacy Scale as a measure of self-efficacy in brain injury by comparing it with other measures of self-efficacy, the GSE, and PROMIS self-efficacy.

DETAILED DESCRIPTION:
Brain injury (BI) can be a devastating experience for many survivors, resulting in chronic difficulties in social, emotional, and physical functioning (Landau & Hissett, 2008). Emotional and neurobehavioral challenges of those with brain injuries often have a direct relationship with their overall rehabilitation outcome. In order to provide patients and caregivers greater support and teach adaptive coping strategies, researchers designed and studied a coping skills group specifically for brain injury survivors and their caregivers at the Rehabilitation Hospital of Indiana (RHI) called the Brain Injury Coping Skills group (BICS). BICS is a 12-session (one session per week), manualized, cognitive-behavioral treatment group designed to provide support, coping skills, and psychoeducation aimed to improve perceived self-efficacy (PSE) and emotional functioning.

Perceived self-efficacy (PSE) is the belief or confidence in one's ability to deal with the challenges related to a specific situation (e.g., brain injury). PSE has been found to be strongly linked to social participation, increased positive regard toward the caregiving role, and was found to be the greatest contributing factor to predicting life satisfaction. Multiple human functions including thought patterns, decisions, motivations, and resiliency are regulated by self-efficacy. PSE also predicts whether an individual can adapt successfully in stressful situations. Cicerone and Azulay found that the greatest contribution to predicting life satisfaction was the person's PSE for managing their cognitive challenges.

Various self-efficacy measures exist. The General Self-Efficacy Scale (GSE) assesses general self-efficacy of the general adult population and adolescents over the age of 12. Additionally, the Patient-Reported Outcomes Measurement Information System (PROMIS) General Self-Efficacy questionnaire that measures an individual's ability to manage various situations, problems, and events, focusing on general life events, as well as social interactions and emotions.

Self-efficacy has been linked with more positive and successful outcomes for brain injury survivors. While low PSE often leads to feelings of depression, anxiety, and avoidance, high self-efficacy often allows points to feelings of more control over one's environment, as well as having a more outward focus on a task, rather than dwelling on themselves and their problems/difficulties. Benight & Bandura noted that self-efficacy is often a predictor in the ability for trauma-survivors to manage their past traumatic experiences. For instance, in combat veterans diagnosed with PTSD, the implementation of self-efficacy exercises reduced stress and anxiety; therefore, these veterans were better able to manage more stressful situations.

Brain injury survivors and their caregivers face unique challenges after the injury, often experiencing difficulties with coping; therefore, it is important that these survivors and their caregivers have positive perceived self-efficacy for better treatment outcomes. Seeing this as a need, the authors of BICS developed the Brain Injury Self-Efficacy Scale which measures perceived self-efficacy in survivors of brain injury and their caregivers. This measure targets this specific population, as they face these unique challenges involving the brain injury (e.g., coping with their injury, and understanding and explaining their injury). The BI Self-Efficacy Scale provided insight to the needs of BI survivors and their caregivers involving self-efficacy; however, it is necessary to validate this measure in order for it to be evidence-based for other survivors of brain injury.

The purpose of this study is to validate the Brain Injury Self-Efficacy Scale as a measure of self-efficacy in brain injury by comparing it with other measures of self-efficacy, the GSE, and PROMIS self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* persons with a history of brain injury (e.g., Traumatic Brain Injury) or acquired BI such as stroke, hypoxia, ruptured aneurysm, or metabolic encephalopathy)
* age 18 and older
* able to speak English fluently.

Exclusion Criteria:

- present with receptive/expressive aphasia preventing them from comprehending the questions or responding appropriately

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are survivors of traumatic or acquired brain injury who are coming into RHI for neuropsychological testing.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Brain Injury Self-Efficacy Scale (BICS-Q) | Baseline
  This measures assesses perceived self-efficacy (PSE) regarding a person's brain injury. The scale ranges from 0 (Not at all confident) to 4 (Extremely confident). This measure provides a total score in which higher scores mean greater self-efficacy.

SECONDARY OUTCOMES:
Patient-reported Outcome Measurement Information System (PROMIS): Self-efficacy for managing symptoms | Baseline
  This measures a person's confidence in managing one's daily activities, emotions, medications/treatments, social interactions, and symptoms. Participants rate how confident they feel about various statements, rating them from 1 (I am not confident at all) to 5 (I am very confident). Higher scores mean higher reported self-efficacy for managing their symptoms.
The General Self-Efficacy Scale (GSE) | Baseline
  This measures assesses general self-efficacy of the general adult population and adolescents over the age of 12. Participants respond to each statement by determining how true it is to their life, using the following scale: Not true at all (1), Hardly true (2), Moderately true (3), Exactly true (4). Scores are totaled and the higher the score, the greater self-efficacy the individual reports.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Hospital of Indiana, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No